CLINICAL TRIAL: NCT00264602
Title: Real-Time Image Guided Lymphatic Mapping and Nodal Targeting in Lung Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Beth Israel Deaconess Medical Center (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Yolonda Colson, MD, PhD, Principal Investigator, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 05-219
Record Dates: First submitted 2005-12-12; First posted 2005-12-13 (Estimated); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer
Keywords: Lymphatic mapping; nodal targeting; indocyanine green; near infrared imaging
MeSH Terms: conditions — Lung Neoplasms | interventions — Indocyanine Green; Sentinel Lymph Node Biopsy

STUDY DESIGN:
Masking Description: There is no masking in this study. All study subjects will receive the same intervention.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Near Infrared Imaging (Experimental): The intervention to be administered is indocyanine green dye.
  Interventions: Drug: Near Infrared Imaging

INTERVENTIONS:
Drug: Near Infrared Imaging — Dye injected into or around tumor at the time of surgery
  Other Names: Indocyanine Green; Sentinel Lymph Node

SUMMARY:
The primary purpose of this study is to determine if we can identify the first lymph node that drains from the tumor, and thus would be the most likely site for metastatic disease, and remove it for analysis to improve the ability to detect tumor in this node and to remove this additional site that potentially contains tumor cells.

DETAILED DESCRIPTION:
* This study is designed to determine the feasibility, safety amd dosing for indocyanine green and near-infrared fluorescent light in order to maximize the near infrared-guided detection of tumor-specific sentinel lymph nodes during the routine surgery for early stage lung cancer when the tumor and nearby lymph nodes are removed.
* At the time of surgery, the indocyanine dye will be injected into or around the patient's tumor. We are using a dose approximately 10,000 times lower than previously approved for injection in the blood. After a few minutes, the surgeon will remove the lymph nodes near the tumor, as is standard for lung surgery, and we will look at these lymph nodes with near-infrared fluorescence.
* The "filtered" near-infrared light causes the indocyanine green dye to fluoresce so that the surgeon can identify the lymph nodes most likely to contain tumor cells. If the lymph node is not found in the group of nodes usually removed, we will use the near-infrared light to look near the tumor for the sentinel lymph nodes and guide the surgeon so that the sentinel nodes can be removed and studied. The surgeon will then continue with the operation and remove the tumor. The lymph nodes are processed for special analysis tailored to finding metastasis in sentinel lymph nodes.
* Since the first question of this study is to determine the smallest dose of indocyanine green that can be used safely for near-infrared detection of the lymph nodes, not all subjects will receive the same dose. The most any person will receive is 1/3 of a teaspoon.
* A five year observation period begins following the operation during which surgeons and physicians will examine the patient and order certain studies to look for evidence of regrowth of the tumor.

ELIGIBILITY:
Inclusion Criteria:

* Suspected or histologically documented new non-small cell carcinoma that have agreed to undergo a thoracotomy for segmentectomy, lobectomy, bilobectomy or pneumonectomy as recommended by their thoracic surgeon for treatment
* Surgically resectable lung cancer
* N2 lymph nodes negative on PET scan or mediastinoscopy
* Age > or equal to 18 years of age
* Men, women of non-child bearing age or women with a negative pregnancy test

Exclusion Criteria:

* Patient does not want to undergo subsequent surgical resection
* Medical condition such as uncontrolled infection or cardiac disease that, i the opinion of the treating surgeon, makes resection unreasonably hazardous for the patient.
* T4 or N2 disease
* Pre-operative spirometry that suggests they cannot undergo resection of their primary tumor by segmentectomy, lobectomy, bilobectomy, or pneumonectomy
* Iodide or seafood allergy
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2009-02-18 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and efficacy of near-infrared technology to guide therapeutic sentinel lymph node dissection in patients with lung cancer. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Yolonda L. Colson, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No